CLINICAL TRIAL: NCT03785288
Title: A Randomized Phase III Trial of Two Standard Dose Fractionation Regimes for Adjuvant Vaginal Brachytherapy in Early Stage Endometrial Cancer
Brief Title: Vaginal Cuff Brachytherapy Fractionation Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kara Romano, MD (Other)
Responsible Party: Sponsor-Investigator, Kara Romano, MD, Principle Investigator-MD Radiation Oncology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20163
Record Dates: First submitted 2018-11-15; First posted 2018-12-24 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will compare two standard of care treatments: HDR vaginal brachytherapy 3 fractions of 7Gy to HDR vaginal brachytherapy 6 fractions of 4Gy for early stage endometrial cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A: 3 treatments of 7Gy (Active Comparator): Arm A: accepted randomization to HDR vaginal brachytherapy in 3 treatments (fractions) of 7Gy for a total dose of 21gy
  Interventions: Radiation: HDR vaginal brachytherapy
- ARM B: 6 treatment of 4Gy (Active Comparator): Arm B: accepted randomization to HDR vaginal brachytherapy 6 treatments (fractions) of 4Gy for a total does of 24gy
  Interventions: Radiation: HDR vaginal brachytherapy
- ARM AB: 6 treatment of 4Gy (Active Comparator): Arm AB: initially randomized to ARM A but wanted to switch to ARM B treatment of HDR vaginal brachytherapy 6 treatments (fractions) of 4Gy for a total does of 24gy
  Interventions: Radiation: HDR vaginal brachytherapy
- ARM BA: 3 treatments of 7Gy (Active Comparator): initially randomized to ARM B but wanted to switch to ARM A of HDR vaginal brachytherapy in 3 treatments (fractions) of 7Gy for a total dose of 21gy
  Interventions: Radiation: HDR vaginal brachytherapy

INTERVENTIONS:
Radiation: HDR vaginal brachytherapy — HDR vaginal brachytherapy 7 Gy in 3 fractions or HDR vaginal brachytherapy 4 Gy in 6 fractions

SUMMARY:
The purpose of this study is to see the effects of two different standard of care treatments of endometrial cancer on sexual dysfunction. This study will compare two standard of care treatments: HDR (high dose radiation) vaginal brachytherapy 3 fractions of 7 Gy to HDR vaginal brachytherapy 6 fractions of 4Gy for early stage endometrial cancer.

DETAILED DESCRIPTION:
Patients are randomized to HDR vaginal brachytherapy 7 Gy in 3 fractions prescribed at 5mm. Radiation delivered 4-12 weeks after surgery OR HDR vaginal brachytherapy 4Gy in 6 fractions prescribed at the cylinder surface. Patients have the option to request to decline their randomization and switch to the alternate treatment ARM if they prefer.

Radiation delivered 4-12 weeks after surgery. Participants in all Arms will receive standard vaginal dilator for use after treatment (to promote healing). 3 month, 1 year and 2 year follow up assessments are performed.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide written informed consent and to comply with the study protocol as judged by the investigator.
* Surgery consisted of Total Abdominal or Laparoscopic Hysterectomy and Bilateral Salpingo Oophorectomy (TH-BSO) with or without lymph node dissection.
* Subject must have FIGO Stage I-II (grade 1-3) pathologically proven (histologic) endometrioid cancer, including all subtypes. Serous, clear cell, and carcinosarcoma histologic pathologies are allowed.
* Subjects must have no measurable disease after surgery.
* ECOG Performance Status of 0-2
* Age ≥ 18 years
* Subject must have a life expectancy ≥ 12 months

Exclusion Criteria:

* Disease of more advanced stage (FIGO stage III-IV) or disease for which adjuvant external beam radiation therapy or chemotherapy is indicated
* Patients with a history of prior pelvic radiation therapy or if additional pelvic radiation therapy is planned
* Subjects who have not recovered from side effects of agents administered more than 4 weeks prior to the on-study date
* Subjects that require > 14 weeks between surgery and initiation of radiation therapy on study unless the subject is receiving chemotherapy. Subjects receiving chemotherapy may have radiation therapy initiated within 6 months after surgery.

  * Subjects who do not meet this criteria may still be eligible. The UVA Coordinating Center and Overall Study PI will review each case and inform the site of the approval decision.
* Subjects who are receiving any investigational agents or have had any investigational agent within the 30 days prior to the on-study date
* Subject is unable or unwilling to participate in a study-related procedure
* Pregnant and breastfeeding women are excluded from this study
* Subject is a prisoner
* A serious uncontrolled medical disorder that in the opinion of the Investigator would impair the ability of the subject to receive protocol therapy.
* Subjects with a history of evidence upon physical examination of central nervous system disease including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (stroke), transient ischemic attack, or subarachnoid hemorrhage within six months of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | 1 year
  Using the FSFI, compare patient reported sexual dysfunction at 1 year after completion of treatment
Preference Option Randomized Design (PORD) | 1 year
  Assessing the comparative effectiveness of receiving HDR vaginal brachytherapy on Arm B or Arm A for early stage endometrial cancer.

SECONDARY OUTCOMES:
Vaginal Length Measurement | 1 year
  Using vaginal dilator compare patient vaginal measurement 1 year after completion of treatment
Vaginal Length Measurement | 2 years
  Using vaginal dilator compare patient vaginal measurement 2 years after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kara Romano, MD, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - University of Maryland Medical Center (UMMC), Baltimore, Maryland
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Virginia, Charlottesville, Virginia